CLINICAL TRIAL: NCT05815264
Title: A Randomized, Blind, Parallel Controlled Phase I Clinical Trial to Evaluate the Safety and Preliminary Immunogenicity of 23-valent Pneumococcal Polysaccharide Vaccine in Healthy Population Aged 2 Years and Older
Brief Title: Clinical Trial of 23-valent Pneumococcal Polysaccharide Vaccine in Healthy Chinese Population Aged 2 Years and Above
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017L04947-1
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental group aged 18-59 years (Experimental): Subjects in the age group 18-59 years received 1 dose of 0.5 mL 23-valent pneumococcal polysaccharide vaccine
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Control group aged 18-59 years (Active Comparator): Subjects in the age group 18-59 years received 1 dose of 0.5 mL pneumococcal vaccine polyvalent
  Interventions: Biological: pneumococcal vaccine polyvalent
- Experimental group aged ≥60 years (Experimental): Subjects in the age group ≥60 years received 1 dose of 0.5 mL 23-valent pneumococcal polysaccharide vaccine
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Control group aged ≥60 years (Active Comparator): Subjects in the age group ≥60 years received 1 dose of 0.5 mL pneumococcal vaccine polyvalent
  Interventions: Biological: pneumococcal vaccine polyvalent
- Experimental group aged 2-17 years (Experimental): Subjects in the age group 2-17 years received 1 dose of 0.5 mL 23-valent pneumococcal polysaccharide vaccine
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Control group aged 2-17 years (Active Comparator): Subjects in the age group 2-17 years received 1 dose of 0.5 mL pneumococcal vaccine polyvalent
  Interventions: Biological: pneumococcal vaccine polyvalent

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — This vaccine（0.5ml） is produced by Ab&b Biotechnology Co., Ltd.JS. Subjects will receive one dose of 23-valent pneumococcal polysaccharide vaccine administered by intramuscular injection.
  Arms: Experimental group aged 18-59 years; Experimental group aged 2-17 years; Experimental group aged ≥60 years
Biological: pneumococcal vaccine polyvalent — This vaccine（0.5ml） is produced by Merck Sharp & Dohme Corp. Subjects will receive one dose of pneumococcal vaccine polyvalent administered by intramuscular injection.
  Arms: Control group aged 18-59 years; Control group aged 2-17 years; Control group aged ≥60 years

SUMMARY:
The group aged 18-59 years old, the group ≥60 years old, and the group aged 2-17 years old were successively assigned to the group. Subjects in each age group were randomly vaccinated with 1 dose of experimental vaccine or control vaccine in a ratio of 1:1, with 48 people in each group receiving each dose. After the safety assessment was conducted on the 8th day after the first dose, the next age group could be enrolled only if the preliminary safety assessment results met the protocol requirements. When each age group is enrolled, laboratory index screening can be conducted 3 days in advance (the validity period of laboratory index detection results is 3 days). The progression of age groups is as follows:

Group 18-59 years old (48 people: 1 dose) → Group ≥60 years old (48 people: 1 dose) → Group 2-17 years old (48 people: 1 dose)

Safety observation: All subjects were observed on site for 30 minutes after vaccination, abnormal laboratory indicators (blood biochemistry, blood routine) of all subjects were observed on day 4 after vaccination, and adverse events of all subjects within 0-7 days were actively followed up by the researchers, and subjects were instructed to record the body temperature measured every day and adverse events (if they occurred) in the diary card. All subjects continued to observe adverse events within 8-28 days and made relevant records. All subjects were required to continue follow-up for SAE status up to 6 months after basic immunization.

Immunogenicity observation: Blood samples were collected before and 28 days after vaccination, and serum antibodies were detected by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* ≥2 years old healthy population;
* Subjects and/or guardians or trustees voluntarily signed informed consent forms and could comply with the requirements of the clinical trial protocol;
* Had not received any pneumonia vaccine in the last 5 years；
* Note: Healthy people do not include the following conditions: ① congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.; ② History of epilepsy and mental illness; ③ Patients with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune diseases; Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases; ⑤ serious liver and kidney diseases, malignant tumors, all kinds of acute diseases or in the acute phase of chronic disease; Adults have diabetes, severe cardiovascular disease, and high blood pressure (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) that cannot be controlled by medication.

Exclusion Criteria:

* Armpit temperature >37.0℃ before inoculation;
* Family history of seizures or convulsions, epilepsy, and mental illness;
* People with a progressive neurological disorder or a history of Guillain-Barre syndrome;
* The patients with clinically significant abnormalities in blood biochemistry and routine blood tests were tested before vaccination；
* People who received immunoenhancement or suppressant therapy within 3 months (continuous oral or intravenous infusion for more than 14 days);
* History of abnormal coagulation function (such as deficiency of coagulation factor, coagulation disease);
* Primary and secondary immunocompromised individuals (thyroid, pancreas, liver, spleen excision history, or need treatment for thyroid disease within the last 12 months);
* History of severe allergic reactions to vaccinations;
* Allergy to any component of the investigational vaccine;
* Have received live attenuated vaccine within 14 days; Other vaccines received within 7 days;
* Participating in or planning to participate in other clinical trials;
* Women of childbearing age are lactating, pregnant or planning to become pregnant in the near future;
* The investigator determined that other conditions were not suitable for participation in the clinical trial.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Incidence of any adverse event within 30 minutes after vaccination. | Within 30 minutes of vaccination
  Incidence of any adverse event within 30 minutes after vaccination.
The incidence of abnormal indicators of blood biochemistry and blood routine on the 4th day after vaccination | Within 4 days of vaccination
  The incidence of abnormal indicators of blood biochemistry and blood routine on the 4th day after vaccination
Incidence of any adverse event within 0-7 days after vaccination. | Within 0-7 days of vaccination
  Incidence of any adverse event within 0-7 days after vaccination.
Incidence of any adverse event within 8-28 days after vaccination. | Within 8-28 days of vaccination
  Incidence of any adverse event within 8-28 days after vaccination.
Incidence of any serious adverse event within 6 months after vaccination. | Within 6 months of vaccination
  Incidence of any serious adverse event within 6 months after vaccination.

SECONDARY OUTCOMES:
Serum IgG antibody seroconversion rate of subjects 28 days after vaccination. | At 28 days after vaccination
  Serum IgG antibody seroconversion rate of subjects 28 days after vaccination.
Serum IgG antibody GMC of subjects 28 days after vaccination. | At 28 days after vaccination
  Serum IgG antibody GMC of subjects 28 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Qi County Center for Disease Control and Prevention, Hebi, Henan, China

IPD SHARING:
Plan to Share IPD: No